CLINICAL TRIAL: NCT01585272
Title: A 52-week, Prospective, Multi-center, Open-label Study to Assess the Tolerability of Rivastigmine Before and After Switching From Oral Formulation to Transdermal Patch in Patients With Alzheimer's Dementia in a Controlled Titration Schedule
Brief Title: Tolerability of Rivastigmine Before and After Switching From Oral Formulation to Transdermal Patch in Alzheimer's Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DTW04
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Alzheimer's Dementia
Keywords: Alzheimer's dementia, AD
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rivastigmine (Experimental): Eligible patients, who are under rivastigmine capsule 3 mg b.i.d. treatment for 4 weeks before Visit 2, will be recruited, followed by treatment switch from oral capsule to transdermal patch for 48 weeks maintenance treatment.
  Interventions: Drug: ENA713

INTERVENTIONS:
Drug: ENA713
  Other Names: Rivastigmine

SUMMARY:
This phase IIIb study is intended to implement a consistent treatment way for switching to Exelon transdermal patch from oral formulation of rivastigmine to stress the importance of (1) advantages of transdermal patch over conventional oral therapies: smooth drug delivery with reduced side effects;(2) encourage treatment compliance in the Alzheimer's dementia setting.

This study is a single-arm, treatment-switched design. Eligible patients, who are under Exelon capsule 3 mg b.i.d. treatment for 4 weeks before Visit 2, will be recruited, followed by treatment switch from oral capsule to patch for 48 weeks maintenance treatment. During the maintenance period, the treatment will be initiated with Exelon Patch 4.6 mg/24 hours (Exelon Patch 5 cm^2) for the first 24 weeks and the dose will be escalated to Exelon Patch 9.5 mg/24 hours (Exelon Patch 10 cm^2) for another 24 weeks if well tolerated. Visits to assess safety are scheduled at baseline, 3 days, 1 week and 2 weeks after the first treatment switch, every 4 weeks until Week 40, and at the end of study (Week 52). The assessment to address the primary objective will focus on the safety of treatment switching (Week 0~28); however the safety assessment will be performed during the whole study period.

ELIGIBILITY:
Inclusion Criteria:

* With diagnosis of mild to moderate Alzheimer's disease.
* Mini-Mental Status Examination score of 10-26 within 3 months before starting oral rivastigmine treatment.
* A clinical diagnosis of probable AD according to NINCDS/ADRDA criteria. The brain scan (magnetic resonance imaging (MRI) or computed tomography (CT) used for establishing that these criteria are met must have been available on the source document within one year prior to study participation.
* Patients who are currently taking or planned to receive Exelon 3 mg capsule twice-daily treatment.
* Written informed consent must be obtained before any assessment is performed.
* If female, must be surgically sterile or at least one year post-menopausal.
* Sufficient education to read, write, and communicate effectively.
* Capable of complying with the requirements of the study

Exclusion Criteria:

* Any advanced, severe or unstable disease that could interfere with study evaluation or completion or put patient at special risk.
* Any medical or neurological condition other than AD that could explain the patient's dementia (e.g., abnormal thyroid function tests, Vitamin B12 or folate deficiency, posttraumatic conditions, Huntington's disease, Parkinson's disease, syphilis).
* Active uncontrolled peptic ulceration, or gastrointestinal bleeding, within the previous 3 months prior to visit 1.
* A current diagnosis of active, uncontrolled seizure disorder.
* A history within the past year or current diagnosis of cerebrovascular disease (e.g., stroke, transient ischemic attacks, aneurysms).
* Bradycardia (< 50 beats per minute), sick sinus syndrome, conduction deficits (S-A block, second or third degree A-V block)
* Severe or unstable cardiovascular disease.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes, or other components of the formulation.
* Current diagnosis of a systemic active skin disorder or lesion that would prevent accurate assessment of the adhesion and skin irritation potential of the patch.
* Previous lack of efficacy with cholinesterase inhibitors.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases. Patients with history of malignancy yet have been treated and defined as complete remission for more than 5 years are not excluded from study participation.
* Pregnant or nursing (lactating) women.
* Concurrently treated with succinylcholine, similar neuromuscular blocking agents or cholinergic agonists such as bethanechol 2 weeks before the start of study drug and during the treatment period.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Taiwan (4):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients receiving Exelon patch 5 cm^2 were more than those receiving Exelon capsule for 4 weeks as least, because some patients had interrupted Exelon capsule for few days in the middle of 4-week Exelon capsule treatment, but still switched to Exelon patch 5 cm2
Period: Overall Study
Arm/Group | Rivastigmine
Started | 121
Safety Set | 102 (Subjects received 3 mg bid Exelon caps for more than 4 weeks & used at least 1 dose of Exelon patch.)
Exelon Patch 5 cm2 | 114
Exelon Patch 10 cm2 | 96
Completed | 82
Not Completed | 39
Not completed — Adverse Event | 22
Not completed — Protocol Violation | 7
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | Rivastigmine
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.8 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events, Serious Adverse Events, and Death
Description: The overall rate of adverse events reported from initiation through the first 28-week treatment period
Time Frame: Baseline through week 28
Population: Safety population: All enrolled subjects who received 3 mg b.i.d Exelon capsule for more than 4 weeks and used at least one dose of Exelon patch therapy.
Measure: Number; unit: Participants
Arm/Group | Rivastigmine
Number analyzed (Participants) | 102
Participants
  Patients with at least one SAEs | 16
  Patients with at least one AE | 94
  Death | 0

2. Secondary Outcome: Change From Baseline in Mini-Mental Status Examination (MMSE)
Description: The changes in Mini-Mental Status Examination (MMSE) of patients with Alzheimer's disease treated with Exelon 5 cm^2 Patch at Week 28 and Exelon 10 cm2 Patch at Week 52 versus baseline, the treatment-switching day at Week 4. MMSE is a multi-item instrument that examines orientation, registration, attention, calculation, recall, visuospatial ability and language. The total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline. The assessments will be conducted at Visit 1, 2, 8, 11 and 17 (screening, Week 4 (baseline), 16, 28 and 52).
Time Frame: Baselin, week 16, 28 and 52
Population: ITT population: All enrolled subjects who received 3 mg b.i.d Exelon capsule orally for 4 weeks and at least one dose of Exelon patch therapy
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Rivastigmine
Number analyzed (Participants) | 102
Score
  Week 16 (n=90) | -0.1 (2.62)
  Week 28 (n=82) | 0.1 (2.62)
  Week 52 (n=93) | -1.0 (3.48)

3. Secondary Outcome: Change From Baseline in Alzheimer Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)
Description: The changes in Alzheimer Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) of patients with Alzheimer's disease treated with Exelon 5 cm^2 Patch at Week 28 and Exelon 10 cm^2 Patch at Week 52 versus baseline, the treatment-switching day at Week 4. ADAS-Cog has been used as the major cognitive measure of anti-dementia drugs. The total score range is 0 to 70 points, with higher scores indicating greater cognitive impairment. The assessments will be conducted at Visit, 2, 8, 11 and 17 (Week 4 (baseline), 16, 28 and 52).
Time Frame: Baseline, week 16, 28 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Rivastigmine
Number analyzed (Participants) | 102
Score
  Week 16 (n=90) | 0.0 (4.92)
  Week 28 (n=82) | 0.4 (5.20)
  Week 52 (n=93) | 0.8 (7.37)

4. Secondary Outcome: The Discontinuation Rate Due to the Treatment Switching From Oral Capsule to Rivastigmine Patch Treatment
Description: The discontinuation rate due to the treatment switching from oral capsule to patch treatment. For patients who discontinue earlier due to intolerance of patch treatment, the proportion will be analyzed. Both the discontinuation rate of 5 cm2 and 10 cm^2 patch therapy will be presented.
Time Frame: Baseline through week 52
Population: Of the patients treated, N=121, number of patients analyzied were those who received 5cm patch (n=114) and those who received 10cm patch (n=96)
Measure: Number; unit: Participants
Arm/Group | Rivastigmine
Number analyzed (Participants) | 114
Participants
  Exelon patch 5 cm 2:Week 4 - Week 28 | 18
  Exelon patch 10 cm 2: Week 28 - Week 52 | 14

5. Secondary Outcome: Percentage of Patients Successfully Titrated to Rivastigmine Patch 10 cm^2
Description: The percentage of patients successfully titrated to rivastigmine patch 10 cm2
Time Frame: Baseline through week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivastigmine
Number analyzed (Participants) | 102
Percentage of participants | 85.3

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Rivastigmine
Serious Adverse Events (participants affected / at risk) | 16/102
Other Adverse Events (participants affected / at risk) | 83/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine (N=102)
Cardiac failure chronic (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Arthritis infective (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pyuria (Infections and infestations) | 1
Tertiary syphilis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Open fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine (N=102)
Cataract (Eye disorders) | 3
Dry eye (Eye disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 6
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 11
Application site erosion (General disorders) | 3
Application site erythema (General disorders) | 18
Application site pruritus (General disorders) | 34
Application site rash (General disorders) | 14
Chest discomfort (General disorders) | 3
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 6
Periodontitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 5
Weight decreased (Investigations) | 28
Decreased appetite (Metabolism and nutrition disorders) | 12
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Dizziness (Nervous system disorders) | 24
Headache (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 4
Irritability (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 3
Papule (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.